CLINICAL TRIAL: NCT05502198
Title: A Rapid, Non-invasive, Clinical Surveillance for CachExia, Sarcopenia, Portal Hypertension and Hepatocellular Carcinoma in End-Stage Liver Disease
Brief Title: Relevance of Sarcopenia in Advanced Liver Disease
Acronym: ACCESS-ESLD
Status: Recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Amra Medical AB (Industry)
Responsible Party: Principal Investigator, Mattias Ekstedt, Associate Professor, Linkoeping University
Other Study IDs: 2020-07215
Record Dates: First submitted 2022-02-15; First posted 2022-08-16 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Liver Cirrhosis; Hepatocellular Carcinoma; Sarcopenia; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Sarcopenia; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with established liver cirrhosis, or end-stage liver disease (ESLD), are at high risk of developing liver cancer (hepatic carcinoma; HCC), portal hypertension, and sarcopenia, all which lead to significant morbidity and mortality. In this patient group the annual incidence of HCC is c. 2-8% and these patients are therefore included in ultrasound HCC screening programs every 6 months.

In this study, the investigators are aiming to assess sarcopenia, clinically significant portal hypertension (CSPH), and HCC with a single short magnetic resonance (MR) examination. A neck-to-knee MRI-examination will be acquired to derive body composition profile (BCP) measurements including visceral and abdominal subcutaneous adipose tissue (VAT and ASAT), thigh fat free muscle volume (FFMV) and muscle fat infiltration (MFI), as well as liver fat (PDFF), spleen volume, and liver stiffness. Images will be further processed by AMRA Medical AB. AMRA's solution includes FFMV in the context of virtual control groups (VCG; using AMRA's vast database) and MFI. Furthermore, the spleen volume will be used to monitor the development of portal hypertension and explored together with other BCP variables in relation to hepatic decompensation events. HCC screening will be performed using so-called abbreviated MRI (AMRI), which consists of time series of contrast-enhanced T1-weighted images. The AMRI images will be read by an experienced radiologist. In the literature the sensitivity of AMRI to detect HCC is above 80%, with a specificity of c. 95%, compared to ultrasound sensitivity of 60%.

In treating ESLD there is a desire of physicians to be able to predict future decompensation events in order to initiate treatment to prolong survival. Moreover, the ability to assess processes of sarcopenia in the patient would be highly valuable for clinical practice due its severe clinical impact. Finally, ultrasound-based HCC screening has poor diagnostic performance and a MR-based screening approach would significantly improve treatment outcome as more treatable and earlier HCC may be identified.

DETAILED DESCRIPTION:
150 patients with established or probable liver cirrhosis at the Department of Gastroenterology and Hepatology at Linköping University Hospital, as well as collaborating hospitals; District Hospital in Eksjö and County Hospital in Jönköping, will be included in the study. The study includes four visits every six months (in patients with LI-RADS 3 five visits will be performed); each patient participates actively in the study during a time period of approximately 24 months. All study visits are scheduled in conjunction with clinical routine visits.

During each study visit the following is performed:

* A detailed clinical work-up
* Assessment of medical history or changes in health status since last visit
* FibroScan
* Magnetic resonance (MR) examination
* Comprehensive blood panels and blood samples for research
* Muscle function and mobility assessments (SPPB and hand grip strength).
* Quality of life assessment (EQ-5D-5L, QLDQ-cirrhosis and SHS-liver).
* Hepatic encephalopathy assessment (ANT test).
* Assessment of the development of symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Established or probable liver cirrhosis according to clinical practice at the Department of Gastroenterology and Hepatology at Linköping University Hospital. This is not by necessity biopsy verified, it can be different criteria such as FibroScan, symptoms, biopsy, and radiology.
2. Age ≥18 years
3. Written informed consent from the participant

Exclusion Criteria:

1. Contraindications for MRI
2. Subjects suffering from primary sclerosing cholangitis (PSC)
3. Subjects diagnosed with Hepatic carcinoma (HCC)
4. Previous liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients with established or probable liver cirrhosis at the Department of Gastroenterology and Hepatology at Linköping University Hospital as well as collaborating hospitals; District Hospital in Eksjö and County Hospital in Jönköping, will be included in the study. All etiologies of cirrhosis will be included except patients with primary sclerosing cholangitis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Body composition (FFMVvcg) | Baseline
  FFMVvcg is the thigh fat-free muscle volume in the context of virtual controls which effectively measures the deviation from expected thigh fat-free muscle volume normalized to height squared using sex and BMI matched virtual control groups.
Body composition (FFMVvcg) | 6 months
  FFMVvcg is the thigh fat-free muscle volume in the context of virtual controls which effectively measures the deviation from expected thigh fat-free muscle volume normalized to height squared using sex and BMI matched virtual control groups.
Body composition (FFMVvcg) | 1 year
  FFMVvcg is the thigh fat-free muscle volume in the context of virtual controls which effectively measures the deviation from expected thigh fat-free muscle volume normalized to height squared using sex and BMI matched virtual control groups.
Body composition (FFMVvcg) | 18 months
  FFMVvcg is the thigh fat-free muscle volume in the context of virtual controls which effectively measures the deviation from expected thigh fat-free muscle volume normalized to height squared using sex and BMI matched virtual control groups.
Change from baseline Body composition (FFMVvcg) | 6 months
  FFMVvcg is the thigh fat-free muscle volume in the context of virtual controls which effectively measures the deviation from expected thigh fat-free muscle volume normalized to height squared using sex and BMI matched virtual control groups.
Change from 6 months Body composition (FFMVvcg) | 1 year
  FFMVvcg is the thigh fat-free muscle volume in the context of virtual controls which effectively measures the deviation from expected thigh fat-free muscle volume normalized to height squared using sex and BMI matched virtual control groups.
Change from 1 year Body composition (FFMVvcg) | 18 months
  FFMVvcg is the thigh fat-free muscle volume in the context of virtual controls which effectively measures the deviation from expected thigh fat-free muscle volume normalized to height squared using sex and BMI matched virtual control groups.
Muscle fat infiltration (%) [MFI] | Baseline
  MFI is a measure, using MR, of percentage of fat infiltration in the muscles (%).
Muscle fat infiltration (%) [MFI] | 6 months
  MFI is a measure, using MR, of percentage of fat infiltration in the muscles (%).
Muscle fat infiltration (%) [MFI] | 1 year
  MFI is a measure, using MR, of percentage of fat infiltration in the muscles (%).
Muscle fat infiltration (%) [MFI] | 18 months
  MFI is a measure, using MR, of percentage of fat infiltration in the muscles (%).
Change from baseline Muscle fat infiltration (%) [MFI] | 6 months
  MFI is a measure, using MR, of percentage of fat infiltration in the muscles (%).
Change from 6 months Muscle fat infiltration (%) [MFI] | 1 year
  MFI is a measure, using MR, of percentage of fat infiltration in the muscles (%).
Change from 1 year Muscle fat infiltration (%) [MFI] | 18 months
  MFI is a measure, using MR, of percentage of fat infiltration in the muscles (%).
Presence of previous decompensation | Baseline
  If the patient previously has had ascites, bleeding esophageal varices, or encephalopathy.
New episode of decompensation since baseline | 6 months
  If the patient has had an episode of ascites, bleeding esophageal varices, or encephalopathy.
New episode of decompensation since 6 months | 1 year
  If the patient has had an episode of ascites, bleeding esophageal varices, or encephalopathy.
New episode of decompensation since 1 year | 18 months
  If the patient has had an episode of ascites, bleeding esophageal varices, or encephalopathy.
New episode of decompensation since 18 months | 2 years
  If the patient has had an episode of ascites, bleeding esophageal varices, or encephalopathy.
Hepatocellular carcinoma | Baseline
  Detection of HCC by AMRI
Significant liver lesion | Baseline
  LI-RADS 3-5
Significant liver lesion | 6 months
  LI-RADS 3-5
Significant liver lesion | 1 year
  LI-RADS 3-5
Significant liver lesion | 18 months
  LI-RADS 3-5
Hepatocellular carcinoma | 6 months
  Detection of HCC by AMRI
Hepatocellular carcinoma | 1 year
  Detection of HCC by AMRI
Hepatocellular carcinoma | 18 months
  Detection of HCC by AMRI
Hepatocellular carcinoma | 2 years
  Chart review
Hand grip strength (kg) | Baseline
  Measured at each visit with a hand-grip dynamometer
Hand grip strength (kg) | 6 months
  Measured at each visit with a hand-grip dynamometer
Hand grip strength (kg) | 1 year
  Measured at each visit with a hand-grip dynamometer
Hand grip strength (kg) | 18 months
  Measured at each visit with a hand-grip dynamometer
Muscle function | Baseline
  Measured using the validated Short Physical Performance Battery.
Muscle function | 6 months
  Measured using the validated Short Physical Performance Battery.
Muscle function | 1 year
  Measured using the validated Short Physical Performance Battery.
Muscle function | 18 months
  Measured using the validated Short Physical Performance Battery.
Child-Pugh score | Baseline
  A validated score to assess prognosis in liver cirrhosis. Includes: Albumin, Bilirubin, INR, Ascites, and Encephalopathy
Child-Pugh score | 6 months
  A validated score to assess prognosis in liver cirrhosis. Includes: Albumin, Bilirubin, INR, Ascites, and Encephalopathy
Child-Pugh score | 1 year
  A validated score to assess prognosis in liver cirrhosis. Includes: Albumin, Bilirubin, INR, Ascites, and Encephalopathy
Child-Pugh score | 18 months
  A validated score to assess prognosis in liver cirrhosis. Includes: Albumin, Bilirubin, INR, Ascites, and Encephalopathy
Child-Pugh score | 2 year
  A validated score to assess prognosis in liver cirrhosis. Includes: Albumin, Bilirubin, INR, Ascites, and Encephalopathy
MELD-score | Baseline
  A validated score to assess prognosis in liver cirrhosis. Includes: Creatinine, INR, Bilirubin, and Sodium
MELD-score | 6 months
  A validated score to assess prognosis in liver cirrhosis. Includes: Creatinine, INR, Bilirubin, and Sodium
MELD-score | 1 year
  A validated score to assess prognosis in liver cirrhosis. Includes: Creatinine, INR, Bilirubin, and Sodium
MELD-score | 18 months
  A validated score to assess prognosis in liver cirrhosis. Includes: Creatinine, INR, Bilirubin, and Sodium
MELD-score | 2 years
  A validated score to assess prognosis in liver cirrhosis. Includes: Creatinine, INR, Bilirubin, and Sodium

SECONDARY OUTCOMES:
Death | 6 months
  Chart review
Death | 1 year
  Chart review
Death | 18 months
  Chart review
Death | 2 years
  Chart review
Esophageal varices | Baseline
  Assessed by gastroscopy and captured through chart review.
Development of Esophageal varices | 6 months
  Assessed by gastroscopy and captured through chart review.
Development of Esophageal varices | 1year
  Assessed by gastroscopy and captured through chart review.
Development of Esophageal varices | 18 months
  Assessed by gastroscopy and captured through chart review.
Development of Esophageal varices | 2 years
  Assessed by gastroscopy and captured through chart review.
Liver stiffness by Fibroscan (kPa) | Baseline
  Liver stiffness is a surrogate marker for fibrosis stage, portal hypertension, and a prognostic marker.
Liver stiffness by Fibroscan (kPa) | 6 months
  Liver stiffness is a surrogate marker for fibrosis stage, portal hypertension, and a prognostic marker.
Liver stiffness by Fibroscan (kPa) | 1 year
  Liver stiffness is a surrogate marker for fibrosis stage, portal hypertension, and a prognostic marker.
Liver stiffness by Fibroscan (kPa) | 18 months
  Liver stiffness is a surrogate marker for fibrosis stage, portal hypertension, and a prognostic marker.
Liver stiffness by MRE (kPa) | Baseline
  Liver stiffness is a surrogate marker for fibrosis stage, portal hypertension, and a prognostic marker.
Liver stiffness by MRE (kPa) | 6 months
  Liver stiffness is a surrogate marker for fibrosis stage, portal hypertension, and a prognostic marker.
Liver stiffness by MRE (kPa) | 1 year
  Liver stiffness is a surrogate marker for fibrosis stage, portal hypertension, and a prognostic marker.
Liver stiffness by MRE (kPa) | 18 months
  Liver stiffness is a surrogate marker for fibrosis stage, portal hypertension, and a prognostic marker.
Spleen volume (ml) | Baseline
  A surrogate marker for portal hypertension and measured by MR.
Spleen volume (ml) | 6 months
  A surrogate marker for portal hypertension and measured by MR.
Spleen volume (ml) | 1 year
  A surrogate marker for portal hypertension and measured by MR.
Spleen volume (ml) | 18 months
  A surrogate marker for portal hypertension and measured by MR.
Quality of life (Questionnaire) | Baseline
  EQ-5D-5L
Quality of life (Questionnaire) | 6 months
  EQ-5D-5L
Quality of life (Questionnaire) | 1 year
  EQ-5D-5L
Quality of life (Questionnaire) | 18 months
  EQ-5D-5L
Quality of life (Questionnaire) | Baseline
  Short Health Scale-liver
Quality of life (Questionnaire) | 6 months
  Short Health Scale-liver
Quality of life (Questionnaire) | 1 year
  Short Health Scale-liver
Quality of life (Questionnaire) | 18 months
  Short Health Scale-liver

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Ekstedt, MD, PhD, Principal Investigator — Linkoeping University
Locations (3):
- Sweden (3):
  - Department of Gastroenterology), District Hospital in Eksjö, Eksjö
  - Department of gastroenterology, County Hospital in Jönköping, Jönköping
  - Department of gastroenterology and hepatology, Linköping

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nasr P, Forsgren M, Balkhed W, Jonsson C, Dahlstrom N, Simonsson C, Cai S, Cederborg A, Henriksson M, Stjernman H, Rejler M, Sjogren D, Cedersund G, Bartholoma W, Ryden I, Lundberg P, Kechagias S, Leinhard OD, Ekstedt M. A rapid, non-invasive, clinical surveillance for CachExia, sarcopenia, portal hypertension, and hepatocellular carcinoma in end-stage liver disease: the ACCESS-ESLD study protocol. BMC Gastroenterol. 2023 Dec 21;23(1):454. doi: 10.1186/s12876-023-03093-8. PMID 38129794